CLINICAL TRIAL: NCT03180918
Title: Male Fertility Preservation Using Cryopreservation of Testicular Tissue Before Highly Gonadotoxic Cancer Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gumy-Pause Fabienne (Other)
Responsible Party: Sponsor-Investigator, Gumy-Pause Fabienne, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PB_2016-01378
Record Dates: First submitted 2017-05-31; First posted 2017-06-08 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Childhood Cancer; Fertility Disorders
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- testicular tissue cryopreservation (Experimental)
  Interventions: Procedure: testicular tissue biopsy

INTERVENTIONS:
Procedure: testicular tissue biopsy — testicular tissue biopsy during general anesthesia

SUMMARY:
Background:

Due to the remarkable improvement in treatments these last decades, long term survival can be expected in more than 80% of childhood cancer patients. Unfortunately, cancer treatments can be harmful to the gonads and can affect reproductive and endocrine functions. While loss of fertility is a major concern for most patients, sperm cryopreservation should be offered to all pubertal male patients. For prepubertal boys, only the experimental option of testicular biopsy in order to cryopreserve testicular stem cells can be proposed.

Primary aims

- To cryopreserve testicular tissue of prepubertal patient receiving highly gonadotoxic oncological treatment.

Secondary aims

* To cryopreserve testicular tissue after failure of sperm cryopreservation in pubertal patient with high risk of infertility
* To create a database in order to record clinical and biological follow-up data
* To create a research biobank for future research projects

Multicentric study: HUG, CHUV, UKBB

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal patients aged 3 months and older
* Peri and pubertal patients after failure of sperm cryopreservation
* Patients presenting high risk of infertility because of gonadotoxic treatments (i.e high dose of alkylating agents, testicular irradiation, total body irradiation).
* Multidisciplinary team consensus in favour of proposition to cryopreserve testicular tissue

Exclusion Criteria:

* Patients under the age of 3 months
* Refusal of the patient and/or his parents
* Treatments that are not highly gonadotoxic

Ages: 3 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2100-01 (Estimated); Study Completion 2100-01 (Estimated)

PRIMARY OUTCOMES:
Number of pediatric cancer patient who will undergo testicular tissue cryopreservation for fertility preservation | 0-20 years

SECONDARY OUTCOMES:
Incidence of complications related to the testicular biopsy (safety) | 0-20 years
  The safety will be assessed by recording the number of complications of the procedure (e.g. bleeding, infection, testicular atrophy)
Comparison of biochemical markers | 0-20 years
  Comparison of biochemical markers (e.g., FSH; LH, AMH; Inhibin B, SHBG and testosterone) between patients who undergo testicular biopsy and controls

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Gumy-Pause, Study Chair — University Hospital, Geneva
Locations (3):
- Switzerland (3):
  - UKBB, Basel
  - Geneva University Hospitals, Geneva
  - CHUV, Lausanne